CLINICAL TRIAL: NCT05926947
Title: Evaluation of Two Plant Formulations for the Management of Glycemia on Pre-diabetic Participants
Brief Title: OXXYNEA® GS: Study for Glycaemia Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GLYCOXY
Record Dates: First submitted 2023-04-20; First posted 2023-07-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Prediabetic State; Overweight
MeSH Terms: conditions — Prediabetic State; Overweight

STUDY DESIGN:
Intervention Model Description: Double blind randomized parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum A (Experimental)
  Interventions: Dietary Supplement: Verum A
- Verum B (Experimental)
  Interventions: Dietary Supplement: Verum B
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Verum A — Formulation of polyphenols from olive leaf extract, blackcurrant extract, pomegranate extract, grapefruit extract
  Arms: Verum A
Dietary Supplement: Verum B — Formulation of polyphenols from olive leaf extract, blackcurrant extract, white kidney bean extract, chromium picolinate and Zinc bisglycinate
  Arms: Verum B
Dietary Supplement: Placebo — Micro crystalline cellulose
  Arms: Placebo

SUMMARY:
The aim of this study is to develop a proof of concept establishing a causal relationship between glycemia improvement through combination of polyphenols-rich botanical extracts or polyphenols-rich botanical extracts associated with white kidney bean extract and chromimum picolinate + zinc bisglycinate with chronic supplementation. Chronic glycemia improvement will be assessed by following the evolution of HbA1c, postprandial glucose and insulin kinetics, and questionnaires. The study design is double blinded randomized with 3 arms and 29 volunteers per arm.

ELIGIBILITY:
Inclusion Criteria:

* Fasting Plasma Glucose 75 - 125 mg/dL
* HbA1c: 5.-6.5 %
* Both sexes
* Overweight BMI range (25-30 Kg/m2)
* Age: 20-50 years old

Exclusion Criteria:

* Metabolic/Chronical disease
* Menopausal women
* Being pregnant, breastfeeding or wanting to have a baby
* Former obese with a history of yoyo effect
* Have been involved in a weight loss program in the past 12 months or subjected to weight reduction surgery
* Having started or quit smoking, having a high alcohol consumption
* Have in the past been in a long-term antibiotherapy (1 month or more) and/or a regular antibiotherapy in the past 12 months
* Allergy to olive, blackcurrant, pomegranate, grapefruit, white kidney bean, or corn.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  Evaluation of changes in the glycated haemoglobin measurements in comparison of the 3 groups
Post prandial glycemia | 12 weeks
  Evaluation of changes in acute and chronic glycemia: Changes in the postprandial glucose measurements in comparison of the 3 groups after the standardized breakfast at baseline, 4th, 8th and 12th week.
Post prandial insulemia | 12 weeks
  Evaluation of changes in acute glycemia: Change in postprandial insulin in comparison of the 3 groups after the standardized breakfast at baseline, 4th, 8th and 12th week.

SECONDARY OUTCOMES:
Body weight | 12 weeks
  Change in the body weight measurements in comparison of the 3 groups
Dual-energy X-ray (DEXA) | 12 weeks
  Evaluation of changes in fat mass and lean mass using a Dual-energy X-ray absorptiometry and compare amongst 3 groups
Magnetic resonance imaging (MRI) | 12 weeks
  Evaluation of changes in various fat layers (visceral, subcutaneous and deep subcutaneous) using a MRI and compare amongst 3 groups
Short Form 12 (SF-12) questionnaire | 12 weeks
  Evaluation of changes in responses to SF-12 questionnaire. SF-12 questionnaire is a health related questionnaire with 12 questions. The total score range from 0-100, with higher score indicating better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Alcaraz, Principal Investigator — UCAM (Universidad Catolica San Antonio de Murcia)
Locations (1):
- UCAM Universidad Católica San Antonio de Murcia, Guadalupe, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided